CLINICAL TRIAL: NCT07176052
Title: Expectation, Pain Outcomes, and Analgesic Efficacy Following Oncology Abdominal Surgery: A Cohort Study
Brief Title: Expectation, Pain Outcomes, and Pain Medication Following Oncology Abdominal Surgery: A Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anja Edith Geisler, Head of Research Nursing, Rigshospitalet, Denmark
Other Study IDs: AEG-abdominalpain-2025
Record Dates: First submitted 2025-08-25; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Cancer, Hepatic; Cancer, Esophagus; Cancer, Pancreas
Keywords: Acute pain; patient expectations; Cancer in the upper abdominal; analgesics; patients self-rating
MeSH Terms: conditions — Liver Neoplasms; Esophageal Neoplasms; Pancreatic Neoplasms; Acute Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Surgery, liver: Located in the liver
  Interventions: Procedure: cancer surgery
- Surgery, esophagus or stomach: Located in the esophagus or stomach
  Interventions: Procedure: cancer surgery
- Surgery, pancreas: Located in the pancreas
  Interventions: Procedure: cancer surgery

INTERVENTIONS:
Procedure: cancer surgery — All surgery will be performed at Copenhagen University Hospital, Rigshospitalet, Denmark

SUMMARY:
This study includes participants undergoing major hepatic surgery, surgery in the esophagus or stomach, or major surgery on the pancreas performed at Copenhagen University Hospital, Rigshospitalet. The aims of the study 1: To record patients' level of catastrophizing preoperatively and pain perioperatively, and pain treatment, as well as related side effects. Furthermore, to investigate whether it is possible to assign the task of rating pain scores to the patient.

2. To investigate patients' expectations preoperatively and the fulfillment of these expectations 30 days after, and the development of chronic pain after 6 months. 3. To record patients' pre- and postoperatively rated health and daily quality of recovery during the seven days of admission. Furthermore, patients' symptoms, levels of pain, and use of analgesics will be assessed 30 days and six months after discharge.

DETAILED DESCRIPTION:
This study includes one main study and two sub-studies. The main study and sub-study 1a are both prospective observational cohort studies. Study 1b is a qualitative study that includes semi-structured interviews with the included patients. No formal sample size calculation was performed, as the study method is exploratory.

Location of the study This study will be conducted at the Department of Transplantation and Organ Surgery at Copenhagen University Hospital, Rigshospitalet, Denmark, from October 1, 2025, to October 1, 2026. Study 1b will be performed by phone.

Participants The participants will include patients undergoing major hepatic surgery, surgery in the esophagus or cardia, or major surgery on the pancreas performed at Rigshospitalet.

Inclusion criteria Patients must meet the following criteria to be suitable for inclusion in the study.

Patients > 18 years undergoing elective primary surgical treatment according to the protocol with curative intent. Patients who can read and understand the Danish language.

Exclusion criteria Patients meeting one or more of the following criteria are ineligible for inclusion in this study.

Patients who are cognitively disabled and cannot mentally cooperate with the study design, as assessed by the investigator.

Procedure for patients who withdraw from the trial In accordance with the Declaration of Helsinki 24, patients have the right to withdraw from the study at any time for any reason, but the reason must be recorded in the patient's Case Report Form if the cause is known.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years undergoing elective surgical treatment in the liver, esophagus/cardia, or pancreas, according to the protocol with curative intent.
* Patients who can read and understand the Danish language.

Exclusion Criteria:

• Patients who are cognitively disabled and cannot mentally cooperate with the study design, as assessed by the investigator.

In accordance with the Declaration of Helsinki, patients have the right to withdraw from the study at any time for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone surgery in the pancreas, hepar or esophagus/cardia at Copenhagen University Hospital, Rigshospitalet
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Median use of analgesics and opioids from the day of surgery until day seven after surgery | 7 days
  All analgesics provided from the day of surgery until seven days after surgery, calculated in median/means for the different surgical groups

SECONDARY OUTCOMES:
Patients' preoperative expectations | At inclusion
  Patients' preoperative expectations evaluated by the treatment expectation questionnaire (TEX-Q. The questionnaire contains 15 questions where the patient can rate their expectations from 0 to ten. 0 is no relief, no benefit or no improvement, and ten represents the opposite. Maximum score is 130 indicating very high expectations.
Daily pain measured by the patients | From the day of surgery until the seventh day after surgery
  Patients will be asked to measure pain during rest and mobilisation, and the location of the pain. Pain will be rated by the Numeric Rating Scale from 0 to ten. 0 is no pain and ten is the worst imaginable pain
Fulfillment of patients´ expecations | 30 days after admission
  Explore in which terms the patients´ expectations were fulfilled by interviewing the patients. We will use a semi-structured interview guide for this purpose.
The development of chronic pain | Six months after admission
  We will interview the patients by phone and ask them to rate their pain and if they are still using analgesics. The pain will be rated by the Numeric Rating Scale from 0 to ten. 0 is no pain and ten is the worst imaginable pain. The analgesics will be mapped according to name and frequency used
Postoperative quality of recovery | The day of surgery until the seventh day after surgery
  The patients will be asked to fill out the QoR-15D questionnaire to rate their postoperative quality of recovery. The questionnaire contains 15 questions with a part A which rates every question from 0 indicating at no point to 10 all the time. Part B is the opposite. A high score indicates a good recovery and the score ranges from 0 to 150.
Health-related quality of life | Preoperatively and 30 days and six months after discharge
  The patients will be asked to fill out the questionnaire EQ-5D-5L to measure health-related quality of life. The questionnaire contains five areas; ability to move, personal care, activities, pain and anxiety/depression. Every arera can be rated in five different ways differing from no problems to it is not possible to perform activities, extreme pain or anxiety. Finally the questionnaire includes a scale from 0 indicating the worst health you can imagine to 100 indicating the very best. The patient should place an X on the number indicating the self-evaluated health
Level of Pain Catastrophizing | preoperatively
  The PCS (Pain Catastrophizing Scale) will be used for this purpose. The PCS is a 13-item self-report questionnaire designed to measure catastrophic thinking related to pain. Each item is rated on a 5-point scale: 0: Not at all, 1: To a slight degree, 2: To a moderate degree, 3: To a great degree, 4: All the time. The total PCS score ranges from 0 to 52, with higher scores indicating greater levels of pain catastrophizing. Scores ≥30 are considered to reflect a clinically relevant level of catastrophizing and correspond to the 75th percentile in chronic pain clinic populations. Scores between the 50th and 75th percentile (typically 20-29) indicate moderate risk, while scores above 30 suggest high risk for persistent pain and disability.
Patient's perceived quality of recovery | The day of surgery until day seven after surgery
  The patient's perceived quality of recovery will be monitored using the QoR-15D. The score ranges from 0 to 15025,26. An excellent quality will be considered for numbers from 136-150. Good quality for 122-135. Moderate quality: 90-121; poor quality: 0-89. Health-related quality of life will be collected preoperatively and at 30 days (+/-7 days) postoperatively using the EQ-5D-5L. The EQ-5D-5L uses five domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on five levels: 1. No problems. 2. Slight problems. 3. Moderate problems. 4. Severe problems. 5. Extreme problems (or unable to do).

CONTACTS AND LOCATIONS:
Overall Officials: Anja Geisler, phd, Principal Investigator — Rigshospitalet, Denmark

IPD SHARING:
Plan to Share IPD: No
I do not need to share the IPD with other researchers

REFERENCES:
- [Background] Hanley C, Ladha KS, Clarke HA, Cuthbertson BC, Wijeysundera DN; METS Study Investigators. Association of postoperative complications with persistent post-surgical pain: a multicentre prospective cohort study. Br J Anaesth. 2022 Feb;128(2):311-320. doi: 10.1016/j.bja.2021.10.027. Epub 2021 Dec 3. PMID 34872718
- [Background] Kleif J, Waage J, Christensen KB, Gogenur I. Systematic review of the QoR-15 score, a patient- reported outcome measure measuring quality of recovery after surgery and anaesthesia. Br J Anaesth. 2018 Jan;120(1):28-36. doi: 10.1016/j.bja.2017.11.013. Epub 2017 Nov 22. PMID 29397134
- [Background] Kleif J, Edwards HM, Sort R, Vilandt J, Gogenur I. Translation and validation of the Danish version of the postoperative quality of recovery score QoR-15. Acta Anaesthesiol Scand. 2015 Aug;59(7):912-20. doi: 10.1111/aas.12525. Epub 2015 Apr 13. PMID 25867135
- [Background] Fantola G, Brunaud L, Nguyen-Thi PL, Germain A, Ayav A, Bresler L. Risk factors for postoperative complications in robotic general surgery. Updates Surg. 2017 Mar;69(1):45-54. doi: 10.1007/s13304-016-0398-4. Epub 2016 Sep 30. PMID 27696276
- [Background] Angelica MD, Fong Y. Patient Expectations and Patient-Reported Outcomes. October 2008; 141: 520-9.
- [Background] Hawker GA, Conner-Spady BL, Bohm E, Dunbar MJ, Jones CA, Ravi B, Noseworthy T, Dick D, Powell J, Paul P, Marshall DA; BEST-Knee Study Team. Patients' Preoperative Expectations of Total Knee Arthroplasty and Satisfaction With Outcomes at One Year: A Prospective Cohort Study. Arthritis Rheumatol. 2021 Feb;73(2):223-231. doi: 10.1002/art.41510. Epub 2020 Dec 26. PMID 32892511
- [Background] Filbay SR, Judge A, Delmestri A, Arden NK, Altman D, Beard D, Carr A, Cooper C, Culliford D, Griffin T, Javaid K, Latham J, Murray D, Pinedo-Villanueva R, Price A, Prieto-Alhambra D, Frisaldi E, Shaibani A, Benedetti F, Waljee J, Mcglinn EP, Sears ED, Chung KC, Roine R, Ohinmaa A, Hailey D, Rief W, Shedden-mora MC, Laferton JAC, Auer C, Petrie KJ, Salzmann S, Schedlowski M, Moosdorf R, Younger J, Gandhi V, Hubbard E, Mackey S, Arrow K, Burgoyne LL, Rainville P, Jumma W, Mohamed M, Joseph L, Canby G, Paungmali A, Sitilertpisan P, Pirunsan U, Verbeek J. Evaluating Patients' Expectations From a Novel Patient-Centered Perspective Predicts Knee Arthroplasty Outcome. Pain Ther 2017; 6: 2146-2152.e4.
- [Background] Visser E, Marsman M, van Rossum PSN, Cheong E, Al-Naimi K, van Klei WA, Ruurda JP, van Hillegersberg R. Postoperative pain management after esophagectomy: a systematic review and meta-analysis. Dis Esophagus. 2017 Oct 1;30(10):1-11. doi: 10.1093/dote/dox052. PMID 28859388
- [Background] Pirie K, Traer E, Finniss D, Myles PS, Riedel B. Current approaches to acute postoperative pain management after major abdominal surgery: a narrative review and future directions. Br J Anaesth. 2022 Sep;129(3):378-393. doi: 10.1016/j.bja.2022.05.029. Epub 2022 Jul 6. PMID 35803751
- [Background] Desai N, El-Boghdadly K, Albrecht E. Epidural vs. transversus abdominis plane block for abdominal surgery - a systematic review, meta-analysis and trial sequential analysis. Anaesthesia. 2021 Jan;76(1):101-117. doi: 10.1111/anae.15068. Epub 2020 May 8. PMID 32385856
- [Background] Hemmerling TM. Pain management in abdominal surgery. Langenbecks Arch Surg. 2018 Nov;403(7):791-803. doi: 10.1007/s00423-018-1705-y. Epub 2018 Oct 3. PMID 30284029
- [Background] Gan TJ, Habib AS, Miller TE, White W, Apfelbaum JL. Incidence, patient satisfaction, and perceptions of post-surgical pain: results from a US national survey. Curr Med Res Opin. 2014 Jan;30(1):149-60. doi: 10.1185/03007995.2013.860019. Epub 2013 Nov 15. PMID 24237004
- [Background] Arnold M, Abnet CC, Neale RE, Vignat J, Giovannucci EL, McGlynn KA, Bray F. Global Burden of 5 Major Types of Gastrointestinal Cancer. Gastroenterology. 2020 Jul;159(1):335-349.e15. doi: 10.1053/j.gastro.2020.02.068. Epub 2020 Apr 2. PMID 32247694
- [Background] Deo SVS, Sharma J, Kumar S. GLOBOCAN 2020 Report on Global Cancer Burden: Challenges and Opportunities for Surgical Oncologists. Ann Surg Oncol. 2022 Oct;29(11):6497-6500. doi: 10.1245/s10434-022-12151-6. Epub 2022 Jul 15. PMID 35838905
- [Background] Sullivan R, Alatise OI, Anderson BO, Audisio R, Autier P, Aggarwal A, Balch C, Brennan MF, Dare A, D'Cruz A, Eggermont AM, Fleming K, Gueye SM, Hagander L, Herrera CA, Holmer H, Ilbawi AM, Jarnheimer A, Ji JF, Kingham TP, Liberman J, Leather AJ, Meara JG, Mukhopadhyay S, Murthy SS, Omar S, Parham GP, Pramesh CS, Riviello R, Rodin D, Santini L, Shrikhande SV, Shrime M, Thomas R, Tsunoda AT, van de Velde C, Veronesi U, Vijaykumar DK, Watters D, Wang S, Wu YL, Zeiton M, Purushotham A. Global cancer surgery: delivering safe, affordable, and timely cancer surgery. Lancet Oncol. 2015 Sep;16(11):1193-224. doi: 10.1016/S1470-2045(15)00223-5. PMID 26427363
- [Background] Flam J. PERIOPERATIVE TREATMENT OF GASTRIC CANCER - SHORT REVIEW. 2021; 49: 103-7
- [Background] Arnold M, Ferlay J, van Berge Henegouwen MI, Soerjomataram I. Global burden of oesophageal and gastric cancer by histology and subsite in 2018. Gut. 2020 Sep;69(9):1564-1571. doi: 10.1136/gutjnl-2020-321600. Epub 2020 Jun 30. PMID 32606208